CLINICAL TRIAL: NCT00014430
Title: Phase I Clinical Trial Of Vinorelbine (Navelbine) And Trastuzumab (Herceptin) In Patients With Carcinoma Of The Breast Or Non-Small Cell Lung Cancer And HER-2/NEU Overexpression
Brief Title: Chemotherapy Plus Trastuzumab in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068543; P30CA023108 (NIH); DMS-9904; NCI-G01-1932
Record Dates: First submitted 2001-04-10; First posted 2004-02-16 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2002-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; stage IIIA breast cancer; recurrent breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Vinorelbine

INTERVENTIONS:
Biological: trastuzumab — Trastuzumab (INN; trade name Herceptin) is a monoclonal antibody that interferes with the HER2/neu receptor. Its main use is to treat certain breast cancers.
  The HER receptors are proteins that are embedded in the cell membrane and communicate molecular signals from outside the cell to inside the cell, and turn genes on and off. The HER proteins regulate cell growth, survival, adhesion, migration, and differentiation-functions that are amplified or weakened in cancer cells. In some cancers, notably some breast cancers, HER2 is over-expressed, and causes breast cells to reproduce uncontrollably.
  Other Names: herceptin
Drug: vinorelbine ditartrate — Vinorelbine (trade name Navelbine) is an anti-mitotic chemotherapy drug that is given as a treatment for some types of cancer, including breast cancer and non-small cell lung cancer.
  Other Names: Navelbine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of vinorelbine plus trastuzumab in treating patients who have refractory or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of vinorelbine in combination with trastuzumab (Herceptin) in patients with HER-2/neu overexpressing unresectable or metastatic non-small cell lung cancer (closed to accrual as of 4/16/01) or refractory locally advanced or metastatic breast cancer.
* Determine the pharmacokinetic and pharmacodynamic profiles of this regimen in this patient population.
* Determine the objective response rate of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of vinorelbine.

Patients receive vinorelbine IV over 5-10 minutes on days 1 and 8, and trastuzumab (Herceptin) IV over 30-90 minutes on days 8 and 15 of course 1 and days 1, 8, and 15 of all subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3 to 6 patients receive escalating doses of vinorelbine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 30-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable or metastatic non-small cell lung cancer

  * Stage IIIB or IV (closed to accrual as of 4/16/01) OR
* Histologically confirmed locally advanced breast cancer that has progressed after first-line chemotherapy or metastatic breast cancer
* HER-2/neu overexpression (1+ to 3+)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Menopausal status:

* Not specified

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* ALT no greater than 3 times ULN

Renal:

* Creatinine no greater than 2 times ULN

Cardiovascular:

* No prior or concurrent unstable angina
* No prior symptomatic congestive heart failure
* No myocardial infarction within the past 6 months
* LVEF at least 45% by echocardiogram or MUGA if received prior anthracycline or anthrapyrazole therapy

Other:

* No prior hypersensitivity to trastuzumab, Chinese hamster ovary cell proteins, or any component of these products
* No other medical illness that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior trastuzumab (Herceptin)

Chemotherapy:

* See Disease Characteristics
* No prior vinorelbine

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1999-11; Primary Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Kaufman, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States